CLINICAL TRIAL: NCT06481514
Title: Fetal Reserve Index (FRI) as a Tool for Improving Surveillance Cardiotocography in Labor.
Brief Title: FRI a Method of Reading Cardiotocography (CTG) in Labor
Acronym: FINIS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ID 6566
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Labor Complication
MeSH Terms: conditions — Obstetric Labor Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (FRI) (Active Comparator): The "Fetal Reserve Index" algorithm will be applied to the first group of patients. In in these patients the fetal reserve index will be calculated every 10 minutes.. For patients with abnormal FRI a 40 minute timer will be started within which it will be necessary to exit the "red zone". If such patients will not be able to exit the red zone within 40 minutes, an additional timer will be started of 30 minutes within which the birth will be completed.
  Interventions: Other: Interpretation of the CTG using FRI score
- group B (No FRI) (Active Comparator): The second group of patients will, however, be managed according to the usual protocols internal management.
  Interventions: Other: Classic interpretation of the CTG

INTERVENTIONS:
Other: Interpretation of the CTG using FRI score — At each of the components of the score will be assigned a score of 1 if the variable evaluated is considered normal, 0 if classified as abnormal. To encourage a simplified clinical interpretation of the different scores obtained (score from 1 to 8) they will be classified into 3 risk categories: Score 5-8: green zone, Score 3-4: zone yellow, Score 1-2: red zone. An FRI of 1-2 (red zone) is to be considered as anomalous
  Arms: group A (FRI)
Other: Classic interpretation of the CTG — evaluate the CTG of group B patients according to the usual internal management protocols
  Arms: group B (No FRI)

SUMMARY:
The objective of the study is to investigate the FRI's ability to identify cases requiring urgent intervention which will present an adverse perinatal outcome (respiratory acidosis, metabolic acidosis, Apgar index, etc.) compared to the classical interpretation of CTG.

Patients whose CTG in labor will be considered non-reassuring will be enrolled and randomized into two groups. The "Fetal Reserve Index" algorithm will be applied to the first group of patients.

The second group of patients will, however, be managed according to the usual protocols internal management.

DETAILED DESCRIPTION:
Patients in active labor and diagnosed with category II CTG will be enrolled and randomized into two groups. Full randomization will be performed by Excel software by generating random numbers using the "Randomise (RAND)" function The "Fetal Reserve Index" algorithm will be applied to the first group of patients. In in these patients the fetal reserve index will be calculated every 10 minutes. At each of the components of the score will be assigned a score of 1 if the variable evaluated is considered normal, 0 if classified as abnormal. The different scores obtained (score from 1 to 8) will be classified into 3 risk categories: Score 5-8: green zone, Score 3-4: zone yellow, Score 1-2: red zone. An FRI of 1-2 (red zone) is to be considered as anomalous. For patients with abnormal FRI a 40 minute timer will be started within which it will be necessary to exit the "red zone". If such patients will not be able to exit the red zone within 40 minutes, an additional timer will be started of 30 minutes within which the birth will be completed. The birth will be completed immediately in case of sentinel events (prolonged bradycardia, detachment of placenta, cord prolapse).

The second group of patients will, however, be managed according to the usual protocols internal management.

ELIGIBILITY:
Inclusion Criteria:

* Women in the active phase of labor who presented when they entered the room I delivered a negative admission test (i.e. a normoreactive CTG according to ACOG) and that subsequently present during labor a diagnosis of category II CTG
* Single term pregnancy
* Signature of informed consent

Exclusion criteria

* Failure to sign the informed consent
* Previous caesarean section (TOLAC)
* Twin pregnancy
* Gestational age <37 weeks
* Known genetic/chromosomal syndromes and/or malformations, excluding heart disease without contraindication to vaginal birth

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — the essential criterion is pregnancy
Enrollment: 290 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
number of cases requiring urgent intervention | 12 MONTHS
  number of cases requiring urgent intervention (vaginal operative delivery / urgent cesarean section) identified by the FRI

SECONDARY OUTCOMES:
number of cases that will present a perinatal outcome adverse events | 12 MONTHS
  number of cases that will present a perinatal outcome adverse events (respiratory acidosis, metabolic acidosis, Apgar index, etc.) identified through the application of the FRI compared to the classical interpretation of the CTG.

CONTACTS AND LOCATIONS:
Overall Officials: Angela BOTTA, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy